CLINICAL TRIAL: NCT03061942
Title: Arthroscopic Rotator Cuff Repair With Synovectomy; Prospective Randomized Controlled Study
Brief Title: Arthroscopic Rotator Cuff Repair With Synovectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hyunchul Jo, Associate professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BRM 17-01
Record Dates: First submitted 2017-02-20; First posted 2017-02-23 (Actual); Last update posted 2018-10-31 (Actual); Status verified 2017-09

CONDITIONS: Rotator Cuff Tears
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Synovectomy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional (Active Comparator): Arthroscopic rotator cuff repair without synovectomy
  Interventions: Other: Arthroscopic rotator cuff repair without synovectomy
- Synovectomy (Experimental): Arthroscopic rotator cuff repair with synovectomy
  Interventions: Other: Arthroscopic rotator cuff repair with synovectomy

INTERVENTIONS:
Other: Arthroscopic rotator cuff repair without synovectomy — 30 subjects will undergo conventional arthroscopic rotator cuff repair without synovectomy.
  Arms: Conventional
Other: Arthroscopic rotator cuff repair with synovectomy — 30 subjects will undergo arthroscopic rotator cuff repair with synovectomy. Synovectomy is an operation performed to remove inflamed synovial membrane of a joint. Arthroscopic synovectomy will be performed with the use of a shaver and a cautery device through the portals for arthroscopic rotator cuff repair.
  Arms: Synovectomy

SUMMARY:
The purpose of this study is to assess the effect of synovectomy on clinical outcomes of arthroscopic rotator cuff repair.

ELIGIBILITY:
Inclusion Criteria:

- Patients with a full-thickness rotator cuff tear undergoing arthroscopic rotator cuff repair

Exclusion Criteria:

* History of shoulder surgery
* Acute trauma on affected shoulder
* Chronic dislocation
* Pyogenic infection
* Rotator cuff arthropathy with glenohumeral osteoarthritis and superior migration of the humeral head
* Isolated subscapularis tear
* Psychiatric problems that precluded informed consent
* An inability to read or write
* Other serious issues that precluded participation in the study
* Open surgery
* Rotator cuff tear with worker's compensation claim
* Refuse to participate in the study
* LOM that need brisement force
* Partial-thickness tear with focal full-thickness extension
* Irrepairable rotator cuff tear
* Subjects who, for any reason, are judged by the investigator to be inappropriate for this study, including a subject who had other severe medical condition or laboratory abnormality, or who is unable to communicate or to cooperate with the investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-03-08 (Actual); Primary Completion 2018-10-26 (Actual); Study Completion 2018-10-26 (Actual)

PRIMARY OUTCOMES:
The worst pain VAS(visual analogue scale) | at 3 months after surgery
  A 10-cm scale marked from ''no pain''(0) to ''unbearable pain''(10) was used.

SECONDARY OUTCOMES:
Constant-Murley score | at 3 months after surgery
  The Constant-Murley score (CMS) is a 100-points scale composed of pain (15 points), activities of daily living (20 points), strength (25 points) and range of motion: forward elevation, external rotation, abduction and internal rotation of the shoulder (40 points). The higher the score, the higher the quality of the function.
The average pain VAS(visual analogue scale) | at 3 months after surgery
  The average pain VAS(visual analogue scale) is the mean of the pain VAS at rest, at night, and with movement.

CONTACTS AND LOCATIONS:
Locations (1):
- Joint & Spine Center, SMG-SNU Boramae Medical Center, Department of Orthopedic Surgery, Seoul National University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No